CLINICAL TRIAL: NCT00350844
Title: A Pilot Study of Hydroxyurea for the Treatment of Pulmonary Hypertension in Children and Young Adults With Sickle Cell Disease
Brief Title: Hydroxyurea for Children and Young Adults With Sickle Cell Disease and Pulmonary Hypertension
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Low subject accrual
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Robert I. Liem, MD, Assistant Professor of Pediatics, NU Feinberg School of Medicine, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12735
Record Dates: First submitted 2006-07-10; First posted 2006-07-11 (Estimated); Results first posted 2013-05-08 (Estimated); Last update posted 2019-08-06 (Actual); Status verified 2019-07

CONDITIONS: Sickle Cell Disease; Pulmonary Hypertension
Keywords: Sickle Cell Disease; Pulmonary Hypertension
MeSH Terms: conditions — Anemia, Sickle Cell; Hypertension, Pulmonary | interventions — Hydroxyurea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hydroxyurea (Experimental)
  Interventions: Drug: Hydroxyurea

INTERVENTIONS:
Drug: Hydroxyurea — 20 mg/kg/day and dose escalating every 2 months until maximum tolerated dose.

SUMMARY:
The goal of this study is to test the hypothesis that hydroxyurea is effective for the specific treatment of secondary pulmonary hypertension found on screening in children and young adults with sickle cell disease.

DETAILED DESCRIPTION:
Increasing evidence suggests that pulmonary hypertension, defined by an elevated tricuspid regurgitant jet velocity (TRJV) on echocardiogram, is a major cause of morbidity and mortality in adults with sickle cell disease (SCD). However, both the prevalence and optimal treatment of pulmonary hypertension in children and young adults with SCD are unknown.

We hypothesize that short term therapy with hydroxyurea will decrease TRJV in children and young adults with pulmonary hypertension found on screening. Patients eligible for treatment will have had evidence of pulmonary hypertension on at least 2 screening echocardiograms. Baseline laboratory tests will be obtained and other causes of secondary pulmonary hypertension will be excluded prior to initiation of treatment. Patients will be treated with hydroxyurea according to a standard dose escalation schedule for a total of 12 months. A clinic visit will be required every 2 months and standard screening for toxicity will be performed monthly. There will be an interim analysis of the primary outcome at 6 months following therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age between 10 and 25 years old
* Sickle cell disease with hemoglobin SS, SC or S-B^0 thalassemia confirmed on hemoglobin electrophoresis
* Tricuspid regurgitant jet velocity (TRJV) equal to or greater than 2.5 m/sec on 2 baseline Doppler echocardiograms at least 3 months apart

Exclusion Criteria:

* Patients already being treated with hydroxyurea
* Patients on a chronic transfusion protocol
* Patients with evidence of hepatic (alanine aminotransferase [ALT] equal to or greater than 2 SD above normal) or renal dysfunction (creatinine [Cr] equal to or greater than 2 SD above normal)
* Patients who are pregnant
* Patients with documented causes of severe pulmonary hypertension other than from SCD

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2006-07; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert I Liem, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study is currently closed to patient accrual at all sites due to poor enrollment, including Children's Memorial Hospital, Washington University, Johns Hopkins and the Medical College of Wisconsin. The FDA was notified in 2010, and the IND was removed for this study.
Groups:
- Hydroxyurea: Hydroxyurea : 20 mg/kg/day and dose escalating every 2 months until maximum tolerated dose.
Period: Overall Study
Arm/Group | Hydroxyurea
Started | 6
Completed | 5
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Hydroxyurea
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Tricuspid Regurgitant Jet Velocity
Description: Primary outcome measure was tricuspid regurgitant jet velocity (TRJV) by echocardiogram after 6 and 12 months of hydroxyurea therapy.
Time Frame: 6 and 12 months after HU therapy begins
Population: Study was terminated and 0 participants were analyzed.
Arm/Group | Hydroxyurea
Number analyzed (Participants) | 0

2. Secondary Outcome: Compliance
Description: Secondary outcome measures included compliance; laboratory measures of therapy-related toxicity; laboratory biomarkers for hemolysis, oxidative stress and endothelial injury; and quality of life measures by Child Health Questionnaire (CHQ).
Time Frame: Throughout study
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Hydroxyurea
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

LIMITATIONS AND CAVEATS:
Early termination leading to no data analysis completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes